CLINICAL TRIAL: NCT00626704
Title: A Phase 1b/2 Study of AMG 655 in Combination With Doxorubicin for the First-Line Treatment of Locally Advanced or Metastatic, Unresectable Soft Tissue Sarcoma
Brief Title: Phase 1b/2 Study of AMG 655 With Doxorubicin for the First-Line Treatment of Unresectable Soft Tissue Sarcoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20060324
Record Dates: First submitted 2008-02-14; First posted 2008-02-29 (Estimated); Last update posted 2015-05-25 (Estimated); Status verified 2015-04

CONDITIONS: Locally Advanced or Metastatic, Unresectable Soft Tissue Sarcoma; Sarcoma; Soft Tissue Sarcoma
Keywords: Sarcoma; Soft Tissue Sarcoma; Locally Advanced or Metastatic, Unresectable Soft Tissue Sarcoma; AMG 655; STS; Doxorubicin; Death receptor; TRAIL receptor; Apoptosis
MeSH Terms: conditions — Neoplasm Metastasis; Sarcoma | interventions — conatumumab; Doxorubicin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): AMG 655 + Doxorubicin
  Interventions: Drug: AMG 655; Drug: Doxorubicin
- Arm 2 (Placebo Comparator): Placebo + Doxorubicin
  Interventions: Other: Placebo; Drug: Doxorubicin

INTERVENTIONS:
Drug: AMG 655 — AMG 655 is an investigational, fully human monoclonal agonist antibody that selectively binds to Death Receptor-5 (DR5).
  Other Names: Conatumumab
  Arms: Arm 1
Other: Placebo — Inactive dummy AMG 655 (to maintain blind)
  Arms: Arm 2
Drug: Doxorubicin — Antineoplastic antibiotic obtained from Streptomyces peucetius. It is a hydroxy derivative of Daunorubicin.

SUMMARY:
This phase 1/2, multicenter, randomized, double-blind, placebo-controlled trial is designed to evaluate the efficacy and safety of AMG 655 when combined with doxorubicin compared with doxorubicin alone in subjects with previously untreated, locally advanced or metastatic, unresectable soft tissue sarcoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed soft tissue sarcoma
* Locally advanced, recurrent, or metastatic, unresectable disease
* Measurable disease according to modified RECIST
* ECOG performance status of 0 or 1
* Men or women at least 18 years of age
* Adequate hematological, renal, hepatic, and coagulation function

Exclusion Criteria:

* Prior treatment with anthracyclines
* Uncontrolled cardiovascular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2007-11; Primary Completion 2009-08 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Progression-Free Survival | Length of Study

SECONDARY OUTCOMES:
Objective response rate, time to response, duration of response, clinical benefit rate, overall survival, incidence of adverse events and clinical laboratory abnormalities, and incidence of anti-AMG 655 antibody formation. | Length of Study

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com